CLINICAL TRIAL: NCT01677000
Title: Clinical Priority Program: Bone Infection; Use of a Registry on Infection to Improve Patient Outcomes and Research Efforts
Brief Title: Clinical Priority Program-Bone Infection Registry
Acronym: CPPInfection
Status: Completed | Type: Observational
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Responsible Party: Sponsor
Organization: AO Innovation Translation Center (Other)
Other Study IDs: CPP Infection Registry
Record Dates: First submitted 2012-08-29; First posted 2012-08-31 (Estimated); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Bone Infection; Staphylococcus Aureus
Keywords: bone infection; staphylococcus aureus; registry
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples nasal and wound specimen
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Establish an international registry of over 400 patients with deep infections involving the bone and/or joint from≥20 centers representing all regions of the world with varied hospital and surgeon practice settings to ensure that registry analyses and research reflect typical clinical practice thereby providing optimal guidance for patients, clinicians, and healthcare researchers. Using a data collection platform that minimizes entry burden, collects most information at the time of surgery, and uses Internet technology to minimize data entry. The registry will include:

1. baseline patient attributes;
2. surgical approach, implants and technology;
3. hospital course;
4. surgeon and institutional characteristics;
5. longitudinal patient outcome,
6. post-procedure complications and revisions,
7. serum/tissue/drainage samples.

DETAILED DESCRIPTION:
Establish an international registry with AOCID of over 400 patients with deep infections involving the bone and/or joint from ≥ 20 centers representing all regions of the world with varied hospital and surgeon practice settings to ensure that registry analyses and research reflect typical clinical practice thereby providing optimal guidance for patients, clinicians, and healthcare researchers. Creation of an AOCID Registry for musculoskeletal infection cases will permit better analysis of the causes, contributing factors including patient immune responses, treatments and clinical outcomes of musculoskeletal infections.

* Establish a practice network that includes ≥ 20 geographically distributed centers. These busy practices will be treating patients with varied geographic status to assure balanced representation of diverse patients and practices.
* Establish a Data Coordinating Core team with AOCID using a data collection platform that minimizes entry burden, collects most information at the time of surgery, and uses Internet technology to minimize data entry.

The registry will include:

* baseline patient attributes
* surgical approach, implants and technology
* hospital course
* surgeon and institutional characteristics
* longitudinal patient outcome
* post-procedure complications and revisions
* serum/tissue/drainage samples

  * Establish a Statistical Support team with AOCID to implement cutting-edge statistical techniques including the use of hierarchical generalized linear latent and mixed effects models to address the complex structure and longitudinal nature of registry data. Multivariable predictive models for outcome(s) of infection will be developed.
  * Establish an Outcomes Measurement Team with AOCID and Investigators from the CPP team to advance the science of infection-specific and global patient-reported outcomes to support efficient data collection of web-based, longitudinal data in this registry and future comparative effectiveness research.
  * Develop new assessment tools and conduct research useful to clinical practice. Establish consensus on the definition of treatment failure- characterized as lack of clinically meaningful improvement in infection, pain or physical function following treatment, validate, and refine prediction algorithms for patients at risk for failure.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Confirmed* oxacillin-/methicillin-sensitive Staphylococcus aureus (OSSA/ MSSA) or methicillin resistant Staphylococcus aureus (MRSA) infection involving a long bone (ie, femur, tibia, fibula, humerus, radius, ulna, and clavicle) with one (or a combination) of the following:

  * Osteomyelitis
  * Fracture fixation hardware /prosthetic joint infection
  * Infection around an arthroplasty
* Ability to understand the content of the patient information / informed consent form and to participate in the clinical investigation
* Signed written informed consent * Confirmed either by positive culture from baseline examination or by positive culture from a prior examination of the same surgical site and definitely ongoing infection with Staphylococcus aureus according to the treating surgeon

Exclusion Criteria:

* Patients who cannot give informed consent
* Patients who cannot attend the follow up visits
* Recent history of substance abuse (ie, recreational drugs, alcohol) that would preclude reliable assessment
* Prisoner

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with diagnosis of Staphylococcus aureus bone infection
Sampling Method: Non-Probability Sample
Enrollment: 297 (Actual)
Dates: Start 2012-06; Primary Completion 2018-12-31 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Details on occurence and treatment of bone infection | 1 December 2012

SECONDARY OUTCOMES:
Surgical approach, implants and technology | 01 December 2012
Patient outcome | 01 December 2012
Post-procedure complications and revisions | 01 December 2012

CONTACTS AND LOCATIONS:
Overall Officials: Stephen L Kates, MD, Principal Investigator — University of Richmond
Locations (21):
- United States (5):
  - University of Missouri Health Care, Columbia, Missouri
  - Unity Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Geisinger Health System, Danville, Pennsylvania
  - University of Richmond, Department of Orthopaedic Surgery, Richmond, Virginia
- Hospital Italiano de Buenos Aires, Buenos Aires, Argentina
- Medizinische Universitaetsklinik Innsbruck, Innsbruck, Austria
- Universitair Ziekenhuis Leuven, Leuven, Belgium
- Foothills Medical Centre, Calgary, Alberta, Canada
- China (5):
  - Southwestern Hospital Chongqing, Chongqing, Chongqing Municipality
  - Affiliated Hospital of Zunyi Medical College, Zunyi, Guizhou
  - Beijing University Third Hospital, Beijing
  - Zhejiang Provincial People's Hospital, Hangzhou
  - Queen Mary Hospital, Hong Kong
- Aarhus University Hospital, Aarhus, Denmark
- Germany (3):
  - Berufsgenossenschaftliche Unfallklinik Murnau, Murnau am Staffelsee, Bavaria
  - Justus-Liebig-Universität, Giessen
  - Universitaetsklinikum Regensburg, Regensburg
- Japan (2):
  - Hokkaido University Graduate School of Medicine, Sapporo, Hokkaido
  - Hamawaki Orthopaedic Hospital, Hiroshima
- Universitätsspital Basel, Basel, Canton of Basel-City, Switzerland